CLINICAL TRIAL: NCT03127293
Title: Is Hyperemesis Gravidarum a Risk Factor for Osteoporosis ?
Brief Title: Hyperemesis Gravidarum and Osteoporosis
Status: Completed | Type: Observational
Sponsor: Adana Numune Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Gulsum Uysal, Medical doctor, Adana Numune Training and Research Hospital
Other Study IDs: 2014/435
Record Dates: First submitted 2017-04-15; First posted 2017-04-25 (Actual); Last update posted 2017-04-26 (Actual); Status verified 2017-04

CONDITIONS: Hyperemesis Gravidarum
MeSH Terms: conditions — Hyperemesis Gravidarum

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum and plasma of samples were than seperated and stored at -80 ºC until the assay. Serum phosphorus (P) and calcium (Ca) were measured by Ion selective electrode (ISE) and alkaline phosphatase (ALP) activity was measured by kinetic enzymatic method, with reagents of Beckman Coulter, on an auto-analyser (Olympus AU5400, Beckman Coulter, Inc., U.S.A.). Serum intact parathormone (iPTH) was analyzed by two-site immunoenzymatic method and 25-hidroxy D levels were analyzed by competetive immunoenzymatic method on UniCel DxI 800 Immunoassay System (Beckman Coulter, Inc., U.S.A.).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Hyperemesis Gravidarum group: Blood samples (10 mL) were drawn at the time of DEXA scans in postpartum period
  Interventions: Diagnostic Test: DEXA
- control group: Blood samples (10 mL) were drawn at the time of DEXA scans in postpartum period
  Interventions: Diagnostic Test: DEXA

INTERVENTIONS:
Diagnostic Test: DEXA — Blood samples (10 mL) were drawn at the time of DEXA scans in postpartum period

SUMMARY:
Hyperemesis Gravidarum (HG) is a common disorder for hospitalization in the first trimester of pregnancy and related to protracted vomiting and nausea. It can be accompanied by ketonuria, dehydration and weight loss. Our aim was to investigate osteoporosis in patients with HG. In our study, we investigated osteoporosis in a total of 79 patients (40 HG and 39 control) by means of dual energy x-ray absorptiometry (DEXA) measurements and laboratory parameters related to HG.

DETAILED DESCRIPTION:
In our study, investigators prospectively enrolled gestational-age matched 40 women with history of HG and 39 women with history of healthy pregnancy in postpartum period, in Kayseri Education and Research Hospital, a tertiary teaching hospital in Kayseri, Turkey between january and december 2015. Ethics approval for the study was obtained from Erciyes School of Medicine and written informed consent was acquired from all subjects.

A total of 40 primigravid singleton pregnant patients aged over 18 years diagnosed with hyperemesis gravidarum and treated with intravenous fluids in first trimester were included in our study as HG group. HG was defined and diagnosed according to the criteria such that the pregnant was admitted one or more times for antepartum hospitalization because of protracted vomiting and nausea accompanied by weight loss, disturbance of electrolyte balance, ketonuria, and dehydration. The first hospitalization had occurred before 20 completed weeks of gestation.

Patients in following conditions were excluded from our study:

* Patients with diagnostic confounders such as overt hyperthyroidism, stomach disease, cholelithiasis, or gastroenteritis
* Patients with chronic illness (e.g.Crohn's disease, colitis ulcerosa, chronic liver disease, diabetes, thyroid disfunction, hyperparathyroidism) and multigenerational pregnancies,
* Patients with history of thyroid surgery, calcium and/or hormone producing tumours, systemic lupus erythematodes,
* Patients with eating disorders,
* Patients with usage of steroids, antiepileptic drugs and/or low molecular weight heparin (long term medication known to affect bone metabolism) and also patients with history of steroid usage for fetal lung maturation.
* Patients with history of osteoporosis, bone fracture in young ages in family. The control group consisted of healthy pregnant women. All patients gave birth between 37-40 gestational weeks. History of supplement containing vitamin usage during pregnancy were noted and also the data regarding demographic variables including age, parity, gravida, abortions, vitamin usage in pregnancy and body mass index (BMI) were asked and recorded.

All patients were performed on a standard dual energy x-ray absorptiometry (DEXA, Hologic Discovery Wi S/N 80848) during early postpartum period ( frequently in two days after birth before discharge of patients) by a single technician. Results for bone area, bone mineral density (BMD), bone mineral content (BMC), T and Z scores for lumbar spine (anteroposterior projection at L1-L4) and right hip were recorded. The radiation dose for all of the scans for lumbar spine and right hip were 4.3 µSv, 4.9 µSv, respectively. According to the World Health Organization (WHO) classification system , T-score ≤-2.5 is classified as osteoporosis and T-score between -2.5 and -1 is classified as osteopenia. In deed, a bone mass reduction more than 2.5 standard deviations compared to young adults of the same gender in DEXA scan (T score) is said to be osteoporosis in WHO criteria . Z score is the number of standard deviations above or below the mean for the patient's age, sex, and ethnicity while T score is the number of standard deviations above or below the mean for healthy 30 year old adult of the same sex, and ethnicity .

Biochemical analysis Blood samples (10 mL) were drawn at the time of DEXA scans in postpartum period and collected into ethylenediaminetetraacetate (EDTA) containing sterile tubes and serum separator tubes (SSTs). Samples were centrifugated at 3000 rpm for 10 minutes at room temperature. Serum and plasma of samples were than separated and stored at -80 ºC until the assay. Serum phosphorus (P) and calcium (Ca) were measured by Ion selective electrode (ISE) and alkaline phosphatase (ALP) activity was measured by kinetic enzymatic method, with reagents of Beckman Coulter, on an auto-analyser (Olympus AU5400, Beckman Coulter, Inc., U.S.A.). Serum intact parathormone (iPTH) was analyzed by two-site immunoenzymatic method and 25-hydroxy D levels were analyzed by competitive immunoenzymatic method on UniCel DxI 800 Immunoassay System (Beckman Coulter, Inc., U.S.A.).

Statistical analysis:

The statistical analyses were performed using SPSS for Windows 13.0. Descriptive statistics of all variables were calculated. Some data have been reported as the mean±standard deviation and percentage where necessary. The t-test was performed to compare means between two groups for normally distributed data, and the Mann-Whitney U-test was used for the non-normally distributed data. The χ2-test was used to compare proportions among groups for categorical data. Values of P<0.05 was accepted as statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with hyperemesis gravidarum
* treated with intravenous fluids in first trimester
* primigravid singleton pregnant patients

Exclusion Criteria:

* Patients with diagnostic confounders such as overt hyperthyroidism, stomach disease, cholelithiasis, or gastroenteritis
* Patients with chronic illness (e.g.Crohn's disease, colitis ulcerosa, chronic liver disease, diabetes, thyroid disfunction, hyperparathyroidism) and multigenerational pregnancies,
* Patients with history of thyroid surgery, calcium and/or hormone producing tumours, systemic lupus erythematodes,
* Patients with eating disorders,
* Patients with usage of steroids, antiepileptic drugs and/or low molecular weight heparin (long term medication known to affect bone metabolism) and also patients with history of steroid usage for fetal lung maturation.
* Patients with history of osteoporosis, bone fracture in young ages in family.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: primigravid singleton pregnant patients
Sampling Method: Probability Sample
Enrollment: 79 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2015-12-15 (Actual); Study Completion 2015-12-15 (Actual)

PRIMARY OUTCOMES:
dual energy x-ray absorptiometry (DEXA) | up to 5 minutes
  All patients were performed on a standard dual energy x-ray absorptiometry (DEXA, Hologic Discovery Wi S/N 80848) during early postpartum period ( frequently in two days after birth before discharge of patients) by a single technician to assess osteoporosis. Blood samples include laboratory parameters associated with osteoporosis (Vitamin D, ALP, P, Ca and PTH).

SECONDARY OUTCOMES:
blood tests | up to 5 minutes
  Blood samples (10 mL) were drawn at the time of DEXA scans in postpartum period and collected into ethylenediaminetetraacetate (EDTA) containing sterile tubes and serum separator tubes (SSTs) to assess osteoporosis. Blood samples include laboratory parameters associated with osteoporosis (Vitamin D, ALP, P, Ca and PTH).

CONTACTS AND LOCATIONS:
Overall Officials: Gulsum Uysal, Principal Investigator — Adana Numune Training and Research Hospital, Adana, Turkey

IPD SHARING:
Plan to Share IPD: Yes
if needed.

REFERENCES:
- [Derived] Uysal G, Cagli F, Akkaya H, Nazik H, Karakukcu C, Sutbeyaz S, Yilmaz ES. Hyperemesis gravidarum is not a negative contributing factor for postpartum bone mineral density. J Chin Med Assoc. 2018 Jul;81(7):619-622. doi: 10.1016/j.jcma.2017.10.010. Epub 2018 Feb 3. PMID 29398518